CLINICAL TRIAL: NCT01986452
Title: CPAP Therapie Mit Telemonitoring Bei Obstruktiver Schlafapnoe Und Apoplexie
Brief Title: Telemonitoring of CPAP Therapy in Apoplexy Patients With OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Collaborators: Reinhard Löwenstein-Stiftung (Unknown)
Responsible Party: Principal Investigator, Georg Nilius, Head of Pneumology Department of Helios Clinic Hagen, Institut für Pneumologie Hagen Ambrock eV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StrOSA2013
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: OSA; Apoplexy
Keywords: OSA; Apoplexy; CPAP; adherence; telemonitoring
MeSH Terms: conditions — Stroke | interventions — Palliative Care; Information Motivation Behavioral Skills Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unattended CPAP therapy (Active Comparator): Therapy data will be examined by reading out the CPAP device after 6 months. Patients can obtain help on own request, corresponding to the standard CPAP prescription routine.
  Interventions: Device: CPAP therapy
- Telemonitoring and support (Experimental): CPAP device therapy data will be downloaded by the study site via GSM modules once a week. In case of poor therapy adherence (defined by a minimum average usage of 3h/night over the week) a contact call will be initiated to motivate patients or solve problems identified by telemonitoring. If active home intervention is required, the study site will inform the healthcare provider to visit the patient in a timely manner.
  Interventions: Device: CPAP therapy; Other: Support

INTERVENTIONS:
Device: CPAP therapy
  Other Names: ICON™
Other: Support
  Other Names: Motivation; Telemonitoring; Software Infosmart Web; GSM module
  Arms: Telemonitoring and support

SUMMARY:
Apoplexy patients with OSA are often not receiving a CPAP therapy due to generally poor acceptance and adherence. There is a great potential to significantly improve the treatment and care of these patients in a time economic way by telemonitoring the therapy in home environment.

This study is planned to prove that telephone consultancy and motivation in times of recorded decreasing CPAP therapy usage can improve adherence, neurological function and quality of life.

DETAILED DESCRIPTION:
Eligible patients with confirmed OSA from neurological rehab department of Helios Clinic Hagen Ambrock are asked to join the study. They will be randomly assigned to one of two arms [CPAP with Telemonitoring (MTM) or without Telemonitoring (OTM)] for 6 months of home treatment after hospital discharge. The MTM arm will receive supporting phone calls when the monitored usage time decreases.

ELIGIBILITY:
Inclusion Criteria:

* s/p ACM (Arteria Cerebri Media Insult)
* Diagnosed OSA AHI >15/h
* Barthel Index item 8 > 5 points (or home assistance)
* Life expectancy >6 month
* Capable of giving consent

Exclusion Criteria:

* Already existing ventilatory support (CPAP, NIV etc)
* Central AI >50% baseline
* Central AI >5/h under CPAP therapy
* Drug abuse
* Pregnant or nursing women
* Participation in another clinical trial last 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Adherence to CPAP usage | 6 months
  CPAP device usage time will be readout and compared.

SECONDARY OUTCOMES:
Quality of life | 6 months
  Patients will fill the questionnaire SF-12 Health Survey before starting the therapy and after 6 months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Hagen
Locations (1):
- Helios Klinik Hagen, Hagen, North Rhine-Westphalia, Germany